CLINICAL TRIAL: NCT06230107
Title: Nutritional Therapeutic Intervention in Eating Disorders
Brief Title: The Effects of Nutritional Intervention in Participants With Eating Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Tatiana Palotta Minari, Principal Investigator, Sao Jose do Rio Preto Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70217317.4.0000.5415
Record Dates: First submitted 2023-12-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Eating Disorders; Binge-Eating Disorder; Binge Eating Disorder Associated With Obesity; Eating Behavior; Eating Disorder
Keywords: eating disorders; binge eating disorder; eating behavior; eating disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: quantitative, prospective, longitudinal and experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants diagnosed with Binge Eating Disorder (Experimental): The intervention was divided into 8 individual weekly meetings, guided by Mindful eating session, nutritional educational dynamics, cooking workshop, food sensory analysis and applications of questionnaires
  Interventions: Behavioral: Mindful Eating

INTERVENTIONS:
Behavioral: Mindful Eating — Analyze the impact of Mindful Eating on changes in dietary habits, episodes of binge eating, body image dissatisfaction, quality of life and anthropometric data (weight, BMI and waist circumference) in Participants with obesity and BED.

SUMMARY:
The goal of this clinical trial is to evaluate the effects of nutritional intervention in eating disorders. Participants underwent an intervention without a control group over 8 weeks. This study aims to provide the maximization of nutritional rehabilitation and support changes in the construction of food autonomy, through a food and nutritional intervention.

DETAILED DESCRIPTION:
Analyze the impact of nutritional intervention on changes in dietary habits, episodes of binge eating, body image dissatisfaction, quality of life and anthropometric data (weight, BMI and waist circumference) of participants with BED. This quantitative, prospective, longitudinal and experimental study recruited 82 participants diagnosed with Obesity and BED. The intervention was divided into 8 individual weekly meetings, guided by Mindful eating session, nutritional educational dynamics, cooking workshop, food sensory analysis and applications of questionnaires (Body Image Scale - BSQ; Binge Eating Scale - BES; Quality of Life Scale - WHOQOL BREF). The meetings occurred from October to November 2023.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with BED who are available to participate

Exclusion Criteria:

* individuals without a diagnosis of BED who are available to participate; who cannot attend meetings; with clinical changes; who have difficulty answering the questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Episodes of Binge Eating {Binge Eating Scale (BES} (0 to 48 points)}. | 8 weeks
  Evaluate the impact of nutritional intervention on the variation in the number of binge eating episodes between the 1st and 8th week. Application of the 'Binge Eating Scale (BES) which quantifies the severity of Binge Eating, cognitions, feelings, and behaviors related to the Binge Eating episode, consisting of 16 items in a 4-point Likert format and 62 statements from which the one that best represents the individual's response. Each statement corresponds to a number of points from 0 to 3, ranging from the absence ("0") to the maximum severity ("3") of Binge Eating. The final score is the result of the sum of the points for each item. According to the classification, individuals with a score less than or equal to 17 are classified as "No Binge Eating". Individuals with a score between 18 and 26 are considered to have "Moderate Binge Eating" and those with a score greater than or equal to 27 are classified as "Severe Binge Eating" (minimum 0 points and maximum 48 points).
Body Image Dissatisfaction {Body Shape Questionnaire (BSQ) (34 to 204 points)}. | 8 weeks
  Evaluate the impact of nutritional intervention on the level of body image dissatisfaction between the 1st and 8th week. Application of the Body Image Scale (BSQ) who was measures satisfaction and concern with body shape, consisting of 34 items on a 6-point Likert scale. According to the classification, to be classified as "satisfied with your body shape" is necessary score <111 (minimum 34 points and maximum 204 points).
Quality of Life {Quality of LifeScale WHOQOL BREF) (0 to 100%)}. | 8 weeks
  Evaluate the impact of nutritional intervention on quality of life between the 1st and 8th week. Application of the Quality of Life Scale WHOQOL BREF who was evaluates the quality of life of the patient, comprising 26 Likert-scale questions. This ques-tionnaire is divided into 4 domains - physical, psychological, social, and environmental. According to the classification, the higher the percentage, the better the quality of life (0-100%)
Weight (kg). | 8 weeks
  Evaluate the impact of nutritional intervention on weight (kg) between the 1st and 8th week.
Body Mass Index (kg/m²). | 8 weeks
  Evaluate the impact of nutritional intervention on Body Mass Index [Weight(kg)/height(m)²] between the 1st and 8th week.
Waist circumference (cm). | 8 weeks
  Evaluate the impact of nutritional intervention on waist circumference (cm) between the 1st and 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Palotta Minari, PhD Student, Principal Investigator — State Faculty of Medicine in São José do Rio Preto
Locations (1):
- Tatiana Palotta Minari, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in eating disorders. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact: tatianaminari@gmail.com